CLINICAL TRIAL: NCT00079339
Title: Phase I/II Trial of R115777 and XRT in Pediatric Patients With Newly Diagnosed Non-Disseminated Intrinsic Diffuse Brainstem Gliomas
Brief Title: Tipifarnib and Radiation Therapy in Treating Young Patients With Brainstem Glioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03021; NCI-2012-03021 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PBTC-014 (Other: Pediatric Brain Tumor Consortium); PBTC-014 (Other: CTEP); U01CA081457 (NIH)
Record Dates: First submitted 2004-03-08; First posted 2004-03-10 (Estimated); Results first posted 2010-09-24 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2012-12

CONDITIONS: Untreated Childhood Brain Stem Glioma
MeSH Terms: interventions — Radiotherapy; Radiation; tipifarnib

ARMS (1):
- Treatment (radiation therapy and tipifarnib) (Experimental): PHASE I: Patients undergo radiotherapy 5 days a week for 6 weeks. Beginning 0-2 days before radiotherapy, patients receive oral tipifarnib twice daily until the completion of radiotherapy. Beginning 2 weeks after the completion of radiotherapy, patients receive oral tipifarnib twice daily in weeks 1-3. Treatment repeats every 4 weeks for up to 24 additional courses (total of 26 courses) in the absence of disease progression or unacceptable toxicity.
  PHASE II: Patients undergo radiotherapy and receive tipifarnib at the MTD as in phase I (closed to accrual as of 1/19/06). Treatment continues for up to 24 months (26 courses) in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: radiation therapy; Drug: tipifarnib

INTERVENTIONS:
Radiation: radiation therapy — Undergo radiotherapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Drug: tipifarnib — Given orally
  Other Names: R115777; Zarnestra

SUMMARY:
Tipifarnib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Radiation therapy uses high-energy x-rays to damage tumor cells. Tipifarnib may make tumor cells more sensitive to radiation therapy. Combining tipifarnib with radiation therapy may kill more tumor cells. This phase I/II trial is studying the side effects and best dose of tipifarnib to see how well it works when given together with radiation therapy in treating young patients with newly diagnosed brain stem glioma. (Phase I closed to accrual as of 1/19/06)

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) of R115777 administered concurrently with radiation therapy to pediatric patients with non-disseminated, diffuse, intrinsic brainstem gliomas who are not receiving enzyme-inducing anti-convulsant drugs (EIACD).

II. To assess the efficacy of R115777 treatment in combination with radiation therapy for patients with non-disseminated, diffuse, intrinsic pontine gliomas as measured by progression-free survival and survival distributions.

SECONDARY OBJECTIVES:

I. To characterize toxicities associated with R115777 treatment in combination with and post radiation therapy.

II. To characterize radiographic changes in brainstem gliomas treated with radiation and R115777 using MRI, perfusion and diffusion imaging and PET scans.

OUTLINE: This is a phase I (closed to accrual as of 1/19/06), multicenter, dose-escalation study of tipifarnib followed by a phase II safety and efficacy study.

PHASE I: Patients undergo radiotherapy 5 days a week for 6 weeks. Beginning 0-2 days before radiotherapy, patients receive oral tipifarnib twice daily until the completion of radiotherapy. Beginning 2 weeks after the completion of radiotherapy, patients receive oral tipifarnib twice daily in weeks 1-3. Treatment repeats every 4 weeks for up to 24 additional courses (total of 26 courses) in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of tipifarnib during radiotherapy until the maximum tolerated dose is determined. The MTD is defined as the dose level preceding that at which 2 of 6 patients experience dose-limiting toxicity.

PHASE II: Patients undergo radiotherapy and receive tipifarnib at the MTD as in phase I (closed to accrual as of 1/19/06). Treatment continues for up to 24 months (26 courses) in the absence of disease progression or unacceptable toxicity.

FOLLOW-UP:

Phase I: Participants contributing only to the phase I part are followed for 90 days after completion of therapy. Adverse events that have not resolved within 90 days after stopping treatment will be followed until resolution.

Phase II: Participants in the phase I part treated at the MTD or participants in the phase II part are followed until the earliest of death or three years after starting treatment.

PROJECTED ACCRUAL: A total of 3-55 patients (3-18 patients for phase I [closed to accrual as of 1/19/06] and a total of 40 patients for phase II [including 6 patients treated in the dose-finding portion of phase I (closed to accrual as of 1/19/06)]) will be accrued for this study within 2.3 years.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed non-disseminated intrinsic diffuse brainstem glioma
* Karnofsky performance scale (KPS) (for > 16 yrs of age) or Lansky performance score (LPS) (for =< 16 years of age) => 50 assessed within two weeks prior to registration
* Prior/concurrent therapy:

  * Chemo: No prior therapy allowed
  * Radiation therapy (XRT): No prior therapy allowed
  * Bone Marrow Transplant: None prior
  * Anti-convulsants: Patients receiving EIACDs will not be eligible; however, patients may switch from EIACDs to non-EIACDs and must then be on non-EIACDs for a minimum of 7 days prior to registration
  * Growth factors: Off all colony forming growth factor(s) > 2 weeks prior to registration (G-CSF, GM-CSF, erythropoietin)
* Absolute neutrophil count >= 1,000/mm^3
* Platelets >= 100,000/mm^3 (transfusion independent)
* Hemoglobin >= 8 gm/dL (transfusion independent)
* Serum creatinine that is less than the upper limit of institutional normal for age or GFR > 70 ml/min/1.73m2
* Bilirubin =< 1.5 time upper limit of normal for age
* SGPT (ALT) and SGOT (AST) < 2.5 times institutional upper limit of normal
* Female patients of childbearing potential must have negative serum or urine pregnancy test; patient must not be pregnant or breast-feeding
* Patients of childbearing or child fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while being treated on this study
* Signed informed consent according to institutional guidelines must be obtained

Exclusion Criteria:

* Patients must not have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy; patients must not have any disease that will obscure toxicity or dangerously alter drug metabolism
* Patients with disseminated intrinsic diffuse brainstem glioma
* Patients taking enzyme-inducing anticonvulsant drugs
* Patients with known allergy to topical or systemic imidazoles (e.g., clotrimazole, ketoconazole, miconazole, econazole)
* Patients receiving any other anticancer or experimental drug therapy
* Patients with uncontrolled infection

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 51 (Actual)
Dates: Start 2004-01; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daphne Haas-Kogan, Principal Investigator — Pediatric Brain Tumor Consortium
Locations (1):
- Pediatric Brain Tumor Consortium, Memphis, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants from PBTC member institutions were enrolled on the phase I component between 01/30/2004 and 01/19/2006. The phase II component of the study opened on 06/02/2006 and completed accrual on 12/26/2007.
Groups:
- Tipifarnib 100-mg/m2: Tipifarnib 100 mg/m2 twice a day for 6 weeks concurrent with radiation therapy followed by a two week rest period. Treatment cycles were 4 weeks (maximum tolerated dose (MTD) estimation period - first 8 weeks). Tipifarnib was continued at 200 mg/m2 twice a day, starting at course 3, for 21 days followed by 7 days of rest. Treatment repeats every 4 weeks for up to 24 additional courses.
  Local radiation (RT) was initiated 1-2 days following the first dose of tipifarnib and was administered once daily, five days per week , at 180 cGy/day fractions for six weeks to a total dose of 5580 cGy.
  All participants treated at this dose level were enrolled to the phase I part of the study only.
- Tipifarnib 125-mg/m2: Tipifarnib 125 mg/m2 twice a day for 6 weeks concurrent with radiation therapy followed by a two week rest period. Treatment cycles were 4 weeks (maximum tolerated dose (MTD) estimation period - first 8 weeks). Tipifarnib was continued at 200 mg/m2 twice a day, starting at course 3, for 21 days followed by 7 days of rest. Treatment repeats every 4 weeks for up to 24 additional courses.
  Local radiation (RT) was initiated 1-2 days following the first dose of tipifarnib and was administered once daily, five days per week , at 180 cGy/day fractions for six weeks to a total dose of 5580 cGy.
  The 125 mg/m2 dose level was determined to be the MTD and therefore the recommended phase II dose. Of the 40 participants treated at this dose level, six were enrolled on the phase I part of the study and 34 were enrolled to the phase II.
- Tipifarnib 150-mg/m2: Tipifarnib 150 mg/m2 twice a day for 6 weeks concurrent with radiation therapy followed by a two week rest period. Treatment cycles were 4 weeks (maximum tolerated dose (MTD) estimation period - first 8 weeks). Tipifarnib was continued at 200 mg/m2 twice a day, starting at course 3, for 21 days followed by 7 days of rest. Treatment repeats every 4 weeks for up to 24 additional courses.
  Local radiation (RT) was initiated 1-2 days following the first dose of tipifarnib and was administered once daily, five days per week , at 180 cGy/day fractions for six weeks to a total dose of 5580 cGy.
  All participants treated at this dose level were enrolled to the phase I part of the study only.
Period: Overall Study
Arm/Group | Tipifarnib 100-mg/m2 | Tipifarnib 125-mg/m2 | Tipifarnib 150-mg/m2
Started | 5 | 40 | 6
Enrolled in Phase I | 5 | 6 | 6
Maximum Tolerated Dose (MTD) Estimation | 3 (2 participants enrolled in the phase I part did not complete the 8 week MTD estimation period.) | 6 | 5 (One participant enrolled in the phase I part did not complete the 8 week MTD estimation period.)
Enrolled in Phase II | 0 (Participants treated at the 100 mg/m2 dose level did not participate in the phase II part.) | 40 (This number includes the 6 patients enrolled on the phase I part.) | 0 (Participants treated at the 150 mg/m2 dose level did not participate in the phase II part.)
Completed | 0 | 1 | 0
Not Completed | 5 | 39 | 6
Not completed — Adverse Event | 1 | 7 | 2
Not completed — Death | 1 | 0 | 0
Not completed — Non-compliance | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 4 | 1
Not completed — Disease progression | 3 | 28 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tipifarnib 100-mg/m2 | Tipifarnib 125-mg/m2 | Tipifarnib 150-mg/m2 | Total
Number analyzed (Participants) | 5 | 40 | 6 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 40 | 6 | 51
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 5.87 [4.68 to 8.23] | 5.48 [3.33 to 16.47] | 5.84 [4.55 to 13.75] | 5.72 [3.33 to 16.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 25 | 5 | 31
  Male | 4 | 15 | 1 | 20
Region of Enrollment [Number; unit: participants]
  United States | 5 | 40 | 6 | 51

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in the Phase I Component With Dose-limiting Toxicities (DLTs) Observed During the First 8 Weeks (Courses 1 and 2) of Tipifarnib Therapy
Description: The dose limiting toxicity (DLT) analysis population consists of phase I participants who developed DLT during the maximum tolerated dose (MTD) estimation period (courses 1 and 2) or who completed the MTD estimation period (courses 1 and 2) without DLTs. DLTs observed during courses 1 and 2 were used to estimate the MTD.
Time Frame: Day 1 of tipifarnib therapy to week 8
Population: Per protocol, participants included phase I participants who developed dose-limiting toxicities during the maximum tolerated dose (MTD) estimation period (courses 1 and 2) or who completed the MTD estimation period (courses 1 and 2) without dose-limiting toxicities.
Measure: Number; unit: Participants
Groups:
- Tipifarnib 100-mg/m2: Tipifarnib 100 mg/m2 twice a day for 6 weeks concurrent with radiation therapy followed by a two week rest period. Treatment cycles were 4 weeks (maximum tolerated dose (MTD) estimation period - first 8 weeks). Tipifarnib was continued at 200 mg/m2 twice a day, starting at course 3, for 21 days followed by 7 days of rest. Treatment repeats every 4 weeks for up to 24 additional courses.
  Local radiation (RT) was initiated 1-2 days following the first dose of tipifarnib and was administered once daily, five days per week , at 180 cGy/day fractions for six weeks to a total dose of 5580 cGy.
  All participants treated at this dose level were enrolled to the phase I part of the study.
- Tipifarnib 150-mg/m2: Tipifarnib 150 mg/m2 twice a day for 6 weeks concurrent with radiation therapy followed by a two week rest period. Treatment cycles were 4 weeks (maximum tolerated dose (MTD) estimation period - first 8 weeks). Tipifarnib was continued at 200 mg/m2 twice a day, starting at course 3, for 21 days followed by 7 days of rest. Treatment repeats every 4 weeks for up to 24 additional courses.
  Local radiation (RT) was initiated 1-2 days following the first dose of tipifarnib and was administered once daily, five days per week , at 180 cGy/day fractions for six weeks to a total dose of 5580 cGy.
  All participants treated at this dose level were enrolled to the phase I part of the study.
Arm/Group | Tipifarnib 100-mg/m2 | Tipifarnib 125-mg/m2 | Tipifarnib 150-mg/m2
Number analyzed (Participants) | 3 | 6 | 5
Participants | 0 | 1 | 4

2. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the interval from initiation of treatment to the earliest of disease progression (tumor increase of 25% over baseline tumor measurement; appearance of new lesion(s); or progressive/worsening neurological status) or death for patients who failed, or to the last date of follow up for patients without failure.
Time Frame: Assessed before the first dose of tipifarnib, every 8 weeks for the first 48 weeks, and then every 12 weeks.
Population: Per protocol 40 participants who received at least one dose of tipifarnib were needed for this objective. The analysis population consists of phase I participants treated at the maximum tolerated dose (MTD) and the participants enrolled to the phase II part.
Measure: Median (Full Range); unit: Months
Arm/Group | Tipifarnib 125-mg/m2
Number analyzed (Participants) | 40
Months | 6.8 [.2 to 18.6]

3. Secondary Outcome: Change From Baseline in Perfusion Ratio at Two Weeks After Completion of Radiation
Description: This study attempted to investigate in an exploratory manner the effect of treatment on changes in neuroimaging meaurements. Neuroimaging changes may have some association with outcome (response, survival, etc.). Perfusion values are obtained from magnetic resonance perfusion imaging and were measured at baseline, every 8 weeks for the first 48 weeks, and then every 12 weeks until treatment is discontinued.
Time Frame: Baseline and two weeks post completion of radiation
Population: The analysis population consists of participants, from both the phase I part and the phase II part, treated at any dose level who had a baseline perfusion ratio value and a second perfusion ratio value measured at approximately 8 weeks after starting treatment.
Measure: Median (Full Range); unit: Ratio
Groups:
- Tipifarnib - Any Dose Level: Participants treated at any dose level who had the baseline and on treatment (two weeks post completion of radiation) MRI perfusion scan.
Arm/Group | Tipifarnib - Any Dose Level
Number analyzed (Participants) | 19
Ratio | -.42 [-7.35 to 4.3]

4. Secondary Outcome: Change From Baseline in Diffusion Ratio at Two Weeks After Completion of Radiation.
Description: This study attempted to investigate in an exploratory manner the effect of treatment on changes in neuroimaging meaurements. Neuroimaging changes may have some association with outcome (response, survival, etc.). Diffusion values are obtained from magnetic resonance diffusion imaging and were measured at baseline, every 8 weeks for the first 48 weeks, and then every 12 weeks until treatment is discontinued.
Time Frame: Baseline and two weeks post completion of radiation
Population: The analysis population consists of participants, from both the phase I part and the phase II part, treated at any dose level who had a baseline diffusion ratio value and a second diffusion ratio value measured at approximately 8 weeks after starting treatment.
Measure: Median (Full Range); unit: Ratio
Groups:
- Tipifarnib - All Dose Levels: Participants treated at any dose level who had the baseline and on treatment (two weeks post completion of radiation) MRI diffusion scan.
Arm/Group | Tipifarnib - All Dose Levels
Number analyzed (Participants) | 35
Ratio | -.13 [-1.61 to .93]

5. Secondary Outcome: Change From Baseline in Volume FLAIR at Two Weeks After Completion of Radiation
Description: This study attempted to investigate in an exploratory manner the effect of treatment on changes in various neuroimaging variables. Neuroimaging changes may have some association with outcome (response, survival, etc.). Volume FLAIR is one parameter obtained from standard magnetic resonance imaging (MRI) studies of the brain. Volume FLAIR was obtained at baseline and within two weeks after completion of radiation.
Time Frame: Baseline and two weeks post completion of radiation
Population: The analysis population consists of participants, from both the phase I part and the phase II part, treated at any dose level who had a baseline volume FLAIR value and a second volume FLAIR value measured at approximately 8 weeks after starting treatment.
Measure: Median (Full Range); unit: cubic centimeters
Groups:
- Tipifarnib - All Dose Levels: Participants treated at any dose level who had the baseline and on treatment (two weeks post completion of radiation) MRI scan.
Arm/Group | Tipifarnib - All Dose Levels
Number analyzed (Participants) | 33
cubic centimeters | -12.45 [-29.45 to 7.86]

6. Secondary Outcome: Mean Tumor to Gray Matter Ratio Measured at Baseline
Description: This study attempts to characterize neuroimaging parameters from positron emission tomography. For each patient, the axial image through the tumor containing the maximum activity per pixel corresponding to the highest FluoroDeoxyGlucose (FDG) uptake was identified and a region of interest (ROI) was drawn based on the FDG definition of the tumor. The mean pixel values within the tumor ROI were normalized by those for normal gray matter to provide ratios of tumor/gray matter. Each patient has a mean tumor to gray matter ratio value and the median of these values across patients is reported.
Time Frame: Baseline
Population: The analysis population consists of participants, from both the phase I part and the phase II part, treated at any dose level who had a baseline PET scan.
Measure: Median (Full Range); unit: Ratio
Groups:
- Tipifarnib - All Dose Levels: Participants treated at any dose level who had a baseline positron emission tomography (PET) scan.
Arm/Group | Tipifarnib - All Dose Levels
Number analyzed (Participants) | 14
Ratio | .64 [.42 to 1.17]

7. Secondary Outcome: Mean Tumor to White Matter Ratio Measured at Baseline
Description: This study attempts to characterize neuroimaging parameters from positron emission tomography. For each patient, the axial image through the tumor containing the maximum activity per pixel corresponding to the highest FluoroDeoxyGlucose (FDG) uptake was identified and a region of interest (ROI) was drawn based on the FDG definition of the tumor. The mean pixel values within the tumor ROI were normalized by those for normal white matter to provide ratios of tumor/white matter. Each patient has a mean tumor to white matter ratio value and the median of these values across patients is reported.
Time Frame: Baseline
Population: as for outcome 6
Measure: Median (Full Range); unit: Ratio
Arm/Group | Tipifarnib - All Dose Levels
Number analyzed (Participants) | 14
Ratio | 1.44 [1.17 to 1.91]

ADVERSE EVENTS:
Time Frame: Clinical and laboratory studies to assess adverse events were scheduled pre-treatment, weekly during the first 8 weeks, every 2 weeks for courses 3 -13, and every 12 weeks for courses 14-26. Additional studies were done at the investigator's discretion.
Arm/Group | Tipifarnib 100-mg/m2 | Tipifarnib 125-mg/m2 | Tipifarnib 150-mg/m2
Serious Adverse Events (participants affected / at risk) | 3/5 | 29/40 | 3/6
Other Adverse Events (participants affected / at risk) | 5/5 | 40/40 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tipifarnib 100-mg/m2 (N=5) | Tipifarnib 125-mg/m2 (N=40) | Tipifarnib 150-mg/m2 (N=6)
Lymphopenia (Blood and lymphatic system disorders) | 0 | 13 | 0
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 0 | 2 | 1
Hypertension (Cardiac disorders) | 0 | 1 | 0
Rash: erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 0 | 1 | 0
Hemorrhage, CNS (Nervous system disorders) | 0 | 3 | 0
Hemorrhage, GU (Renal and urinary disorders) | 0 | 1 | 0
Hemorrhage/bleeding associated with surgery, intra-operative or postoperative (Surgical and medical procedures) | 1 | 0 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 0 | 3 | 1 — Blood related
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Infections and infestations) | 0 | 2 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 1 | 0 | 0 — Catheter-related
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 0 | 1 | 0 — Conjunctiva
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 0 | 3 | 0
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 | 2 | 0
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 0 | 2 | 0
Alkalosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 0 | 1 | 0
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 0 | 1 | 0
GGT (gamma-Glutamyl transpeptidase) (Metabolism and nutrition disorders) | 0 | 1 | 0
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 0 | 1 | 0
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 0 | 1 | 0
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 | 1 | 0
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Somnolence/depressed level of consciousness (Psychiatric disorders) | 3 | 4 | 0
Ataxia (incoordination) (Nervous system disorders) | 1 | 3 | 0
Hydrocephalus (Nervous system disorders) | 1 | 3 | 0
Neuropathy: cranial (Nervous system disorders) | 1 | 1 | 0 — CN VI Lateral deviation of eye
Neuropathy: cranial (Nervous system disorders) | 1 | 1 | 0 — CN X Motor-palate; pharynx, larynx
Neuropathy: cranial (Nervous system disorders) | 1 | 1 | 0 — CN IX Motor-pharynx; Sensory-ear, pharynx, tongue
Neuropathy: motor (Nervous system disorders) | 1 | 1 | 0
Seizure (Nervous system disorders) | 0 | 2 | 0
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 1 | 1 | 0
Apnea (Nervous system disorders) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Laryngeal nerve dysfunction (Nervous system disorders) | 0 | 1 | 0
Mood alteration (Psychiatric disorders) | 0 | 1 | 0
Neurology - Other (Specify, __) (Nervous system disorders) | 0 | 1 | 0
Neuropathy: cranial (Nervous system disorders) | 1 | 0 | 0 — CN VIII Hearing and balance
Neuropathy: cranial (Nervous system disorders) | 1 | 0 | 0 — CN VII Motor-face; Sensory-taste
Eyelid dysfunction (Eye disorders) | 0 | 1 | 0
Pain - Kidney (Renal and urinary disorders) | 0 | 1 | 0
Pain - Head/Headache (General disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Obstruction, GU (Renal and urinary disorders) | 0 | 1 | 0 — Ureter
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 0 | 1 | 0
Death not associated with CTCAE term (General disorders) | 2 | 5 | 0 — Disease progression NOS
Death not associated with CTCAE term (General disorders) | 1 | 1 | 0 — Death NOS
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tipifarnib 100-mg/m2 (N=5) | Tipifarnib 125-mg/m2 (N=40) | Tipifarnib 150-mg/m2 (N=6)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 1 | 10 | 3
Lymphopenia (Blood and lymphatic system disorders) | 3 | 29 | 2
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 4 | 25 | 4
Hemoglobin (Blood and lymphatic system disorders) | 1 | 20 | 3
Platelets (Blood and lymphatic system disorders) | 3 | 12 | 3
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2 | 10 | 2
Hypertension (Cardiac disorders) | 0 | 7 | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 | 18 | 3
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 0 | 3 | 1
Weight gain (General disorders) | 1 | 2 | 1
Weight loss (General disorders) | 0 | 3 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 | 15 | 2
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 2 | 7 | 2
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 | 7 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 5 | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 | 5 | 2
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Flushing (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Cushingoid appearance (e.g., moon face, buffalo hump, centripetal obesity, cutaneous striae) (Endocrine disorders) | 2 | 13 | 2
Vomiting (Gastrointestinal disorders) | 3 | 30 | 3
Nausea (Gastrointestinal disorders) | 1 | 17 | 2
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 | 10 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 10 | 1
Anorexia (Gastrointestinal disorders) | 0 | 8 | 3
Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 1 | 7 | 2
Constipation (Gastrointestinal disorders) | 2 | 18 | 4
Hemorrhage, CNS (Nervous system disorders) | 0 | 6 | 0
Hemorrhage, pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 0 | 3 | 0 — External ear (otitis externa)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 1 | 3 | 0 — Middle ear (otitis media)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 1 | 4 | 0 — Mucosa
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 1 | 2 | 0 — Upper airway NOS
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 3 | 22 | 3
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 3 | 16 | 3
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 2 | 17 | 3
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 3 | 11 | 2
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2 | 13 | 1
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 4 | 8 | 3
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 | 12 | 1
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1 | 12 | 1
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 | 10 | 0
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 0 | 8 | 1
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 0 | 7 | 1
GGT (gamma-Glutamyl transpeptidase) (Metabolism and nutrition disorders) | 0 | 5 | 0
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 0 | 4 | 0
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 0 | 4 | 0
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 0 | 3 | 0
Metabolic/Laboratory - Other (Specify, __) (Metabolism and nutrition disorders) | 2 | 1 | 1
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 0 | 3 | 0
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 — Left-sided
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 — Right-sided
Ataxia (incoordination) (Nervous system disorders) | 2 | 29 | 3
Neuropathy: cranial (Nervous system disorders) | 3 | 21 | 2 — CN VI Lateral deviation of eye
Neuropathy: cranial (Nervous system disorders) | 1 | 21 | 3 — CN VII Motor-face; Sensory-taste
Neuropathy: motor (Nervous system disorders) | 1 | 12 | 3
Dizziness (Nervous system disorders) | 0 | 8 | 2
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 1 | 8 | 1
Neuropathy: cranial (Nervous system disorders) | 2 | 6 | 0 — CN X Motor-palate; pharynx, larynx
Mood alteration - Depression (Psychiatric disorders) | 0 | 3 | 1
Neuropathy: cranial (Nervous system disorders) | 2 | 4 | 0 — CN III Pupil, upper eyelid, extra ocular movements
Neuropathy: cranial (Nervous system disorders) | 1 | 5 | 0 — CN IX Motor-pharynx; Sensory-ear, pharynx, tongue
Neuropathy: sensory (Nervous system disorders) | 1 | 4 | 1
Pyramidal tract dysfunction (e.g., increased tone, hyperreflexia, positive Babinski, decreased fine (Nervous system disorders) | 1 | 5 | 0
Somnolence/depressed level of consciousness (Psychiatric disorders) | 1 | 4 | 1
Neuropathy: cranial (Nervous system disorders) | 2 | 3 | 0 — CN XII Motor-tongue
Tremor (Nervous system disorders) | 1 | 4 | 0
Personality/behavioral (Psychiatric disorders) | 0 | 2 | 2
Mood alteration - Agitation (Psychiatric disorders) | 0 | 5 | 1
Neuropathy: cranial (Nervous system disorders) | 0 | 3 | 0 — CN IV Downward, inward movement of eye
Neuropathy: cranial (Nervous system disorders) | 0 | 3 | 0 — CN XI Motor-sternomastoid and trapezius
Neuropathy: cranial (Nervous system disorders) | 0 | 3 | 0 — CN II Vision
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 1 | 13 | 1
Nystagmus (Eye disorders) | 1 | 10 | 0
Vision-blurred vision (Eye disorders) | 1 | 1 | 1
Pain - Head/headache (General disorders) | 2 | 23 | 4
Pain - Abdomen NOS (General disorders) | 1 | 8 | 2
Pain - Extremity-limb (General disorders) | 2 | 5 | 2
Pain - Throat/pharynx/larynx (General disorders) | 0 | 4 | 0
Pain - Back (General disorders) | 0 | 3 | 0
Pain - Middle ear (General disorders) | 0 | 3 | 0
Pain - Eye (General disorders) | 1 | 1 | 1
Pain - Muscle (General disorders) | 0 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 8 | 3
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 | 4 | 1
Incontinence, urinary (Renal and urinary disorders) | 1 | 2 | 0
Urinary frequency/urgency (Renal and urinary disorders) | 0 | 2 | 1
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 3 | 14 | 3
Pain - Stomach (General disorders) | 1 | 1 | 0
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 0 | 1 | 1
Heartburn/dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1
Alkaline phosphatase (Metabolism and nutrition disorders) | 0 | 1 | 1
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 — Lower Extremity
Ocular surface disease (Eye disorders) | 0 | 1 | 1
Vision-photophobia (Eye disorders) | 0 | 1 | 1
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Neuropathy: cranial (Nervous system disorders) | 1 | 1 | 0 — CN V Motor-jaw muscles; Sensory-facial
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 0 | 1 | 1 — Sinusitis NOS
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 0 | 1 | 1 — Urinary tract infection NOS
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 1 | 1 | 0 — Skin infection
Sweating (General disorders) | 0 | 0 | 1
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Febrile neutropenia (fever of unknown origin) (Infections and infestations) | 0 | 0 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 0 | 0 | 1 — Upper aerodigestive NOS
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 0 | 0 | 1 — Bronchitis NOS
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 0 | 0 | 1 — Bladder (urinary)
Infection with unknown ANC (Infections and infestations) | 0 | 0 | 1 — Catheter-related
Opportunistic infection associated with >=Grade 2 Lymphopenia (Infections and infestations) | 0 | 0 | 1
Extremity-lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Extremity-upper (function) (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain - Chest/thorax NOS (General disorders) | 0 | 0 | 1
Pain - Neck (General disorders) | 0 | 0 | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less